CLINICAL TRIAL: NCT07302165
Title: PreParent: Internet-based Digital Tools to Screen for and Prevent Postpartum Depression in Parents-to-be: Identifying and Targeting Cognitive Risk Factors
Brief Title: PreParent: Internet-based Digital Tools to Screen for and Prevent Postpartum Depression in Parents-to-be
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Mental Health Centre Copenhagen, Bispebjerg and Frederiksberg Hospital (Other)
Collaborators: University of Bergen (Other); University of Copenhagen (Other); University of Southern Denmark (Other); Lund University (Other)
Responsible Party: Principal Investigator, Kamilla Woznica Miskowiak, Professor, Mental Health Centre Copenhagen, Bispebjerg and Frederiksberg Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: p-2024-16735
Record Dates: First submitted 2025-12-11; First posted 2025-12-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Post-partum Depression
Keywords: Prevention intervention; Postpartum depression; Digital psychiatry; Online therapy; Risk factors; Pregnancy
MeSH Terms: conditions — Depression, Postpartum

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Online prenatal affective cognitive training (Experimental): Participants in this arm receive a 4-5-week online intervention consisting of 8-9 modules. The program includes psychoeducation on perinatal emotional health and cognitive-affective training exercises designed to reduce risk factors for postpartum depression. All content is completed independently on the online platform.
  Interventions: Behavioral: Online prenatal affective cognitive training
- Care as usual (CAU) (No Intervention): Participants in this arm receive care-as-usual (CAU) provided within the Danish healthcare system. They do not receive access to the online intervention but complete the same assessments and follow-ups as the intervention group.

INTERVENTIONS:
Behavioral: Online prenatal affective cognitive training — Participants receive a 4-5 week online intervention concisting of 8-9 modules. The program includes psychoeducation on perinatal emotional health and cognitive-affective training exercises designed to reduce risk factors for postpartum depression. All content is completed idenpendently on the online platform.
  Arms: Online prenatal affective cognitive training

SUMMARY:
The goal of this randomized controlled study is to evaluate whether an online intervention that combines psychoeducation and affective cognitive training can help prevent postpartum depression in pregnant women and co-parents who have been identified as having risk factors for postpartum depression through an online screening tool. A total of 520 expecting parents will be enrolled in the intervention trial.

Researchers will compare the online intervention to care as usual (CAU) in the Danish healthcare system to determine whether the intervention has a better preventive effect. The study also involves a low-risk comparison group (n = 5250) who will not receive the intervention but will complete the same assessments for background comparisons.

The main question is:

- Does the online intervention reduce the number of mothers who develop postpartum depression during the first six months after birth?

Other questions the study addresses include:

* How severe mothers' depressive symptoms are during the first six weeks postpartum, based on weekly online ratings?
* How do parents report their own stress levels and their infant's development six months after birth?

The study will also explore:

* How many co-parents develop postpartum depression during the first six months postpartum.
* Whether mothers experience additional benefit if their co-parent also completes the intervention.

Participants will:

* Complete a 4-5-week online intervention with 8-9 modules that include psychoeducation and cognitive-affective training.
* Complete online questionnaires and outcome assessments from home.
* Participate in a diagnostic interview by phone after birth.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women in their second or third trimester, or co-parents.
* Age ≥ 18 years.
* Ability to speak and read Danish.
* A cut-off score > 96 on a test of negative cognitive bias (scale 0-100), and/or a score > 23 on the Antenatal Risk Questionnaire (ANRQ).
* Co-parents are categorized as at risk if their partner is identified as having risk factors.

Exclusion Criteria:

* Current or past mental disorders within ICD-10 categories F00-F29 and F60-F69.
* Current substance use.
* EPDS score ≥ 11 for women or ≥ 10 for men, indicating clinically relevant depressive symptoms at baseline.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 520 (Estimated)
Dates: Start 2025-08-30 (Actual); Primary Completion 2027-02-28 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Occurrence of Postpartum Depression in Mothers Assessed at 6 Months Postpartum | 6 months postpartum
  Measured using the Present State Examination (PSE) diagnostic interview at 6 months postpartum to determine whether participants meet criteria for postpartum depression.

SECONDARY OUTCOMES:
Average Severity of Maternal Depressive Symptoms During the First 6 Weeks Postpartum | Weekly assessments from birth to 6 weeks postpartum
  Measured using weekly online ratings on the Edinburgh Postnatal Depression Scale (EPDS). Scores are averaged across the 6-week postpartum period to estimate overall symptom severity.
Self-Reported Parental Stress at 6 Months Postpartum | 6 months postpartum
  Measured using an online questionnaire assessing parental stress levels at 6 months after birth.
Parent-Reported Infant Development at 6 Months Postpartum | 6 months postpartum
  Measured using an online parent-report questionnaire assessing infant developmental functioning at 6 months of age.

OTHER OUTCOMES:
Occurrence of Postpartum Depression in Co-Parents Assessed at 6 Months Postpartum | 6 months postpartum
  Measured using the Present State Examination (PSE) diagnostic interview at 6 months postpartum to determine whether co-parents meet criteria for postpartum depression.
Occurrence of Postpartum Depression in Mothers Whose Co-Parent Also Receives the Intervention | 6 months postpartum
  Exploratory comparison evaluating whether mothers whose co-parent also completes the online intervention show lower occurrence of postpartum depression at 6 months postpartum, compared with mothers whose co-parent does not receive the intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Frederiksberg Hospital, Mental Health Services - Capital Region of Denmark, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] Bjertrup AJ, Kofoed J, Egmose I, Wendelboe K, Southgate V, Vaever MS, Miskowiak KW. Prenatal affective cognitive training to reduce the risk of postpartum depression (PACT): study protocol for a randomized controlled trial. Trials. 2024 Jul 15;25(1):478. doi: 10.1186/s13063-024-08316-1. PMID 39010232
- [Result] Bjertrup AJ, Vaever MS, Miskowiak KW. Prediction of postpartum depression with an online neurocognitive risk screening tool for pregnant women. Eur Neuropsychopharmacol. 2023 Aug;73:36-47. doi: 10.1016/j.euroneuro.2023.04.014. Epub 2023 Apr 27. PMID 37119561
- [Result] Bjertrup AJ, Jensen MB, Schjodt MS, Parsons CE, Kjaerbye-Thygesen A, Mikkelsen RL, Moszkowicz M, Frokjaer VG, Vinberg M, Kessing LV, Vaever MS, Miskowiak KW. Cognitive processing of infant stimuli in pregnant women with and without affective disorders and the association to postpartum depression. Eur Neuropsychopharmacol. 2021 Jan;42:97-109. doi: 10.1016/j.euroneuro.2020.10.006. Epub 2020 Nov 3. PMID 33158668